CLINICAL TRIAL: NCT06494709
Title: Pilot Study of Quantitative Evaluation of Attention to Faces of Patients With Orthognathic Surgery Using Eye-tracking
Brief Title: Quantitative Evaluation of Attention to Faces After Orthognathic Surgery With Eye-tracking
Acronym: OCHIRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Institut Faire Faces (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0146
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Dentofacial Deformities; Orthognathic Surgery; Social Perception; Eye Tracking
Keywords: Dentofacial Deformities; orthognathic surgery; social perception; eye tracking
MeSH Terms: conditions — Dentofacial Deformities | interventions — Moire Topography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: photographs — Standardized photographs presenting 10 control subjects (class I) and patients with dentofacial deformities (10 class II and 10 class III) before and after surgery - from the front and from the side - will be used to form an approximately 10 min video sequence using the Tobii Pro Lab® software (Tobii Pro AB, Danderyd, Sweden). The naive participants will look at the percept during which the faces of the controls and the patients will alternate, with the only instruction being free visual exploration of the percept.
  The fixation duration in the defined areas of interest (eyes, nose, mouth, chin) will be recorded with a Tobii® Pro X3-120 eye-tracking device and the results will be processed with the Tobii Pro Lab® software.

SUMMARY:
Dentofacial deformities refer to morphological anomalies of the jaws. Their development during growth determines the shape of the lower third of the face and the type of dental occlusion. A maxillo-mandibular dysmorphosis associates morphological modification of the face and anomaly of the occlusion. If these anomalies are most often hereditary, they also depend on acquired factors such as swallowing, breathing, sucking or phonation disorders. Angle's classification defines three classes of dental occlusion: class I, when the ratio between the maxillary and mandibular first molars is normal, class II when the upper molar is too far forward, and class III when it is too far back. Class II and III dysmorphoses can result in an alteration of the masticatory function, pain (TMJ, headaches) or sleep apnea. At the same time, they cause patients to experience a decrease in self-esteem, anxiety and social discomfort. Class II and II usually require orthodontic treatment and orthognathic surgery to correctly align the jaws. This surgery has a positive impact on the dental occlusion and the functions concerned, but also on the facial morphology, all of which often leads to an improvement in the patient's quality of life.

Standardized photographs presenting control subjects (class I) and patients (class II and class III) before and after surgery will be included in an approximately 10 min video sequence. Naive participants will look at this sequence during which the faces of the controls and the patients - before and after surgery - will alternate, with the instruction being free visual exploration of the images. The total fixation durations in defined areas of interest (eyes, nose, mouth, chin) will be recorded with an eye tracking device and the results will be processed using a dedicated software.

ELIGIBILITY:
Inclusion Criteria:

* Naïve subject with regard to dentofacial deformities and their management
* Subject with no known facial pathology
* Subject having provided an informed consent
* Subject > 18 years old

Exclusion Criteria:

* Subject familiar with dentofacial deformities and their management (e.g., health professionals in the relevant specialties)
* Subject with known facial pathology (dentofacial deformity or other)
* Subject under guardianship, curators or justice protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Total fixation duration in the "lower third of the face (mouth/chin)" area of interest | one day
  Total fixation duration in the "lower third of the face (mouth/chin)" area of interest, measured in seconds with eye-tracking technique

SECONDARY OUTCOMES:
Total fixation duration in the "eyes" area of interest | one day
  Total fixation duration in the "eyes" area of interest, measured in seconds with eye-tracking technique
Total fixation duration in the "nose"" area of interest | one day
  Total fixation duration in the "nose" area of interest, measured in seconds with eye-tracking technique
Total fixation duration in the eyes", the "nose" and the "lower third of the face (mouth/chin)" areas of interest in patients before orthognathic surgery compared to control subjects. | one day
  Total fixation duration in the eyes", the "nose" and the "lower third of the face (mouth/chin)" areas of interest in patients before orthognathic surgery compared to control subjects.
  measured in seconds with eye-tracking technique
Total fixation duration in the eyes", the "nose" and the "lower third of the face (mouth/chin)" areas of interest in patients after orthognathic surgery compared to control subjects. | one day
  Total fixation duration in the eyes", the "nose" and the "lower third of the face (mouth/chin)" areas of interest in patients after orthognathic surgery compared to control subjects.
  measured in seconds with eye-tracking technique
Total fixation duration in the eyes", the "nose" and the "lower third of the face (mouth/chin)" areas of interest in class II patients before orthognathic surgery compared to class III patients. | one day
  Total fixation duration in the eyes", the "nose" and the "lower third of the face (mouth/chin)" areas of interest in in class II patients before orthognathic surgery compared to class III patients.
  measured in seconds with eye-tracking technique

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens University Hospital, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No